CLINICAL TRIAL: NCT00059436
Title: Mental-effort Effect on Large Muscle Strengthening
Brief Title: Mental Effort and Muscle Strength
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R01HD036725 (NIH)
Record Dates: First submitted 2003-04-25; First posted 2003-04-28 (Estimated); Last update posted 2016-09-26 (Estimated); Status verified 2011-05

CONDITIONS: Aging; Muscle Strength
Keywords: Muscle strengthening; Skeletal muscle Contractions; Rehabilitative exercise

INTERVENTIONS:
Behavioral: Mental effort in muscle strengthening

SUMMARY:
The purpose of this study is to determine the effect of mental effort on improving muscle strength.

DETAILED DESCRIPTION:
Training that involves heavy loads or resistance strengthens muscles. Recent data suggest that substantial voluntary strength gains can be achieved with training involving low resistance and strong mental effort. In contrast, individuals who train with the same low intensity contractions but with low mental effort show no improvement in strength.

This study will evaluate the relationship between mental effort muscle strength improvements by comparing the improvement in muscle strength in participants who have trained with different levels of mental effort. In addition to evaluating muscle strength, this study will also examine the neural mechanisms underlying muscle strength improvements.

Four groups of volunteers (65 years old and over) will participate in a training program directed at elbow-flexor muscles. One group will be trained with an intensity near the level of maximal voluntary contraction (MVC group); a second group will be trained with high mental effort, low muscle intensity contractions (HME group); a third group will be trained with low mental effort, low muscle intensity elbow-flexion contractions (LME group); and the fourth (control) group will not be trained but will participate in the strength tests. Training will be performed every weekday for 12 weeks. Participants will be evaluated by functional MRI (fMRI), EEG-derived motor activity-related cortical potential (MRCP), surface EMG signals, and the MRI T2 relaxation time.

Preliminary analysis of results shows that the HME group gained more than 13% strength, the LME group showed a statistically insignificant 6% change, and the no-practice control group did not show any change in elbow flexor muscle strength. We expect the MVC group to have the highest strength gains among the four groups.

ELIGIBILITY:
Inclusion Criteria

* Healthy individuals free of neurological impairment

Exclusion Criteria

* Already involved in regular physical training
* Neuromuscular disorders
* Medications known to affect neuromuscular system (other than moderate alcohol or caffeine)
* Left-hand dominant

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Dates: Start 1999-10; Primary Completion 2004-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guang H. Yue, Ph.D., Principal Investigator — Cleveland Clinic Foundation, Biomedical Engineering
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States